CLINICAL TRIAL: NCT03863314
Title: Virtual Reality vs Inperson Simulation: A Non-inferiority Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 48883
Record Dates: First submitted 2019-02-28; First posted 2019-03-05 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Work-Related Condition
Keywords: Virtual Reality; Simulation; Workplace

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Person Simulation (Active Comparator): Participants will experience in-person simulations of different workplace scenarios such as medical error and workplace harassment
  Interventions: Other: In-person Simulation
- Virtual Simulation (Experimental): Participants will experience virtual simulations of different workplace scenarios such as medical error and workplace harassment via Virtual Reality headset.
  Interventions: Device: Virtual Simulation

INTERVENTIONS:
Device: Virtual Simulation — Virtual simulation of workplace-related scenarios of pre-recorded videos using the same actors
  Arms: Virtual Simulation
Other: In-person Simulation — In-person simulation of workplace-related scenarios with live actors
  Arms: In-Person Simulation

SUMMARY:
The purpose of this study is to determine if Virtual Reality (VR) can elicit emotional responses that are captured via physiological biometrics such as heart rate variability and skin conductance levels. As a non-inferiority study the investigators anticipate the technologies will elicit an emotional not inferior to those responses of an in-person simulations of workplace scenarios (i.e medical error and workplace harassment).

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* Personnel working or volunteering at Lucile Packard Children's Hospital (LPCH) or Stanford Health Care (SHC) facilities

Exclusion Criteria:

* Patients who do not consent
* Are currently taking beta blockers or other chronotropic heart medication(s)
* Have a history of severe motion sickness
* Currently have nausea
* Currently experiencing seizures
* Are clinically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Respiratory sinus arrhythmia | Throughout duration of simulation, approximately 15 minutes
  Biometric sensors will be placed in strategic locations in order to collect respiratory sinus arrhythmia throughout either in-person or virtual simulation

SECONDARY OUTCOMES:
Skin conductance levels | Throughout duration of simulation, approximately 15 minutes
  Skin conductance levels as measured by electrodermal activity will be collected using biometric sensors throughout either in-person or virtual simulation
Emotional levels | Throughout duration of intervention, two minutes before and after the intervention
  Emotional affect will be self reported via validated scale before and after the intervention.
VR Simulation Questionnaire | Three months post study, approximately 5 minutes
  Participants will be given a questionnaire regarding their virtual or in-person simulation experience and the overall similarity to real-life on a scale from 1-5 (1=Completely Different and 5=Nearly Identical) Example Questions: "How true to real life were the emotions expressed during the scenario?" and "How true to real life was the the clinical environment?"

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States

REFERENCES:
- [Background] Bernardo A. Virtual Reality and Simulation in Neurosurgical Training. World Neurosurg. 2017 Oct;106:1015-1029. doi: 10.1016/j.wneu.2017.06.140. PMID 28985656
- [Background] Kyaw BM, Saxena N, Posadzki P, Vseteckova J, Nikolaou CK, George PP, Divakar U, Masiello I, Kononowicz AA, Zary N, Tudor Car L. Virtual Reality for Health Professions Education: Systematic Review and Meta-Analysis by the Digital Health Education Collaboration. J Med Internet Res. 2019 Jan 22;21(1):e12959. doi: 10.2196/12959. PMID 30668519
- [Background] Fan YC, Wen CY. A Virtual Reality Soldier Simulator with Body Area Networks for Team Training. Sensors (Basel). 2019 Jan 22;19(3):451. doi: 10.3390/s19030451. PMID 30678276